CLINICAL TRIAL: NCT00428636
Title: Study of Early Closure of Temporary Loop Ileostomy After Elective Rectal Resection With Low Pelvic Anastomoses
Brief Title: Early Temporary Stoma Closure After Proctectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM 00154
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Ileostomy
Keywords: ileostomy; rectal resection; proctectomy; stoma closure
MeSH Terms: interventions — Ileostomy

INTERVENTIONS:
Procedure: ileostomy

SUMMARY:
We conducted a prospective randomized study to evaluate the results of early closure of temporary loop ileostomy at eight days in comparison with late closure at two months, after elective rectal resection with low pelvic anastomoses.

DETAILED DESCRIPTION:
The aim of this multicentric prospective randomized study is to compare for patients requiring rectal resection followed by under Douglassienne anastomosis (low colorectal, coloanal, ileoanal) protected by ileostomy, two strategies about delay of ileostomy closing : delayed closing of ileostomy when second hospitalization two months later (classical attitude) ; precocious closing of ileostomy during the same hospitalization (at Day 8 of first operation). All patients aged 18 years or older with disease (carcinoma, inflammatory bowel disease, benign disease) requiring colorectal or rectal resection with low pelvic anastomoses (LPA) (ie low colorectal, coloanal, or ileoanal procedures) were eligible to participate in the study. A water-soluble contrast enema examination through temporary loop ileostomy was performed at day 7. If there were no radiologic signs of contrast leakage, patients were allotted to the group of early closure (EC) or to the group of late closure (LC). The primary end point was the rate of either postoperative death or postoperative complications occurring at 90 days after the first initial procedure.Postoperative complications will be considered present for a patient if one of the following elements is observed during the study : post operative death, anastomotic fistula, postoperative peritonitis ; serious event requiring hospitalization : prolapsus or peristomial eventration, erosive peristomial dermitis, serious wall sepsis, dehydration with hydroelectrolytic disorders, occlusive syndrome.

ELIGIBILITY:
Inclusion Criteria:

* All patients were aged 18 years or older ; there was no upper limit for age.
* All patients with disease (carcinoma, inflammatory bowel disease, benign disease) requiring elective rectal resection with low pelvic anastomosis (ie low colorectal, coloanal, or ileoanal procedures)
* Written informed consent was obtained from all patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2001-05; Study Completion 2005-07

PRIMARY OUTCOMES:
mortality and morbidity rates at three months - The primary end point was the rate of patients with at least one postoperative complications occurring during the first 90 days after the first initial procedure or dying postoperatively

SECONDARY OUTCOMES:
functional results were assessed at 3 and 12 months after the first operation - Quality of life was measured using the Gastrointestinal Quality of Life Index (GICLI)

CONTACTS AND LOCATIONS:
Overall Officials: Yves Panis, Professor, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Hôpital AMBROISE PARE - Service de Chirurgie Digestive, Boulogne-Billancourt, Île-de-France Region
  - Hôpital Cochin - Service de Chirurgie Digestive, Paris, Île-de-France Region
  - Hôpital Lariboisière - Service de Chirurgie Digestive, Paris, Île-de-France Region

REFERENCES:
- [Derived] Alves A, Panis Y, Lelong B, Dousset B, Benoist S, Vicaut E. Randomized clinical trial of early versus delayed temporary stoma closure after proctectomy. Br J Surg. 2008 Jun;95(6):693-8. doi: 10.1002/bjs.6212. PMID 18446781